CLINICAL TRIAL: NCT06283368
Title: Red Blood Cell Distributions (RDW, RDW-CW) and Lymphocyte Monocyte Ratios (LMR) for the Detection of Malignant Thyroid Nodules in the Preoperative Period.
Brief Title: Red Blood Cell Distributions (RDW, RDW-CW) and Lymphocyte Monocyte Ratios (LMR) for the Malignant Thyroid Nodules
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Mehmet Buğra Bozan, Professor, Associate, Kahramanmaras Sutcu Imam University
Other Study IDs: 2021/11-06
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Thyroid Neoplasms Benign; Thyroid Nodule; Thyroid Cancer; Thyroid Diseases
MeSH Terms: conditions — Thyroid Nodule; Thyroid Neoplasms; Thyroid Diseases | interventions — Thyroidectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Benign Thyroid Pathologies: Nodular Goiter Graves Diseases Tocsic Thyroid Nodular Disease
  Interventions: Procedure: Thyroidectomy, Bilaterally Total; Procedure: Thyroidectomy, Unilaterally Total; Procedure: Thyroidectomy, Complementary; Procedure: Thyroidectomy, Near Total
- Thyroid Cancer Cases: Papillary Thyroid Carcinoma Medullary Thyroid Carcinoma Hurthle Cell Carcinoma Anaplastic Thyroid Carcinoma
  Interventions: Procedure: Thyroidectomy, Bilaterally Total; Procedure: Thyroidectomy, Unilaterally Total; Procedure: Thyroidectomy, Complementary; Procedure: Thyroidectomy, Near Total

INTERVENTIONS:
Procedure: Thyroidectomy, Bilaterally Total — Thyroidectomy, Bilaterally Total
Procedure: Thyroidectomy, Unilaterally Total — Thyroidectomy, Unilaterally Total
Procedure: Thyroidectomy, Complementary — Thyroidectomy, Complementary
Procedure: Thyroidectomy, Near Total — Thyroidectomy, Near Total

SUMMARY:
Thyroid surgery is the most common type of surgery among endocrine surgeries. This surgery is performed for patients with suspected malignancy, patients diagnosed with malignancy, and toxic nodular goiter. In addition to vocal cord injury, which is the most important complication of thyroid surgery, hypocalcemia due to hypoparathyroidism and surgical wound complications (such as hematoma, and fistula) can also be observed, and malignancy surgery increases the risk of recurrent laryngeal nerve injury. Therefore, it is important to differentiate these groups using non-invasive methods before surgery.

Tumor-related inflammation is activated as a result of bone marrow and inflammation induced by malignancies. Insufficiently controlled or uncontrolled inflammatory activity may be responsible for malignant transformation. Lymphocyte monocyte ratio and red blood cell distribution are parameters (RDW, RDW-CW) previously studied in terms of cancers.

Our aim in this study is to reveal the RDW, RDW-CW, and LMR calculated from complete blood count parameters in the preoperative period, as an indicator of malignant inflammatory response, in a non-invasive and inexpensive way before surgery or biopsy is performed to distinguish nodular goiter and thyroid malignancy.

DETAILED DESCRIPTION:
Thyroid surgery patients older than 18 who were operated on at the Department of General Surgery of Kahramanmaras Sutcu Imam University between January 2016 and January 2021 for nodular goiter and thyroid malignancy (surgical procedures include bilateral total thyroidectomy, unilateral total thyroidectomy, bilateral subtotal thyroidectomy, unilateral subtotal thyroidectomy, bilateral near total, completion thyroidectomy for recurrent cases). Patients will be evaluated as malignant patients and patients with benign goiter diseases according to the pathology results. Lymphocyte-monocyte ratios will be calculated manually by recording lymphocyte numbers, monocyte numbers, and red blood cell distribution volumes (RDW and RDW-CW) in the routine complete blood count values of the patients in the preoperative period. Patient data will be accessed from the preoperative laboratory and postoperative pathology results recorded in patient epicrisis forms and the computer system.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 age
* Thyroidectomy cases

Exclusion Criteria:

* Younger than 18 age
* Patients with other system malignancies
* Patients with missing data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who need thyroid surgery for the malignant and benign ethiologies
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Determining benign thyroid nodules | 2016-2021
  Determining benign thyroid nodules noninvasively in the preoperative period with complete blood cell parameters
Determining malignant thyroid nodules | 2016-2021
  Determining malignant thyroid nodules noninvasively in the preoperative period with complete blood cell parameters

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bozan MB, Yazar FM, Kale IT, Yuzbasioglu MF, Boran OF, Azak Bozan A. Delta Neutrophil Index and Neutrophil-to-Lymphocyte Ratio in the Differentiation of Thyroid Malignancy and Nodular Goiter. World J Surg. 2021 Feb;45(2):507-514. doi: 10.1007/s00268-020-05822-6. Epub 2020 Oct 16. PMID 33067685
- [Background] Lee F, Yang PS, Chien MN, Lee JJ, Leung CH, Cheng SP. An Increased Neutrophil-to-Lymphocyte Ratio Predicts Incomplete Response to Therapy in Differentiated Thyroid Cancer. Int J Med Sci. 2018 Nov 23;15(14):1757-1763. doi: 10.7150/ijms.28498. eCollection 2018. PMID 30588200
- [Background] Wen W, Wu P, Li J, Wang H, Sun J, Chen H. Predictive values of the selected inflammatory index in elderly patients with papillary thyroid cancer. J Transl Med. 2018 Sep 21;16(1):261. doi: 10.1186/s12967-018-1636-y. PMID 30241494
- [Background] Yaylaci S, Tosun O, Sahin O, Genc AB, Aydin E, Demiral G, Karahalil F, Olt S, Ergenc H, Varim C. Lack of Variation in Inflammatory Hematological Parameters between Benign Nodular Goiter and Papillary Thyroid Cancer. Asian Pac J Cancer Prev. 2016;17(4):2321-3. doi: 10.7314/apjcp.2016.17.4.2321. PMID 27221938